CLINICAL TRIAL: NCT06254261
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase 2 Study Evaluating the Safety, Tolerability, and Efficacy of RAY1225 in Participants With Obesity
Brief Title: A Study of RAY1225 in Participants With Obesity
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Raynovent Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RAY1225-23-02
Record Dates: First submitted 2024-02-03; First posted 2024-02-12 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RAY1225 (cohort 1) (Experimental): Participants received dose1 or dose2 RAY1225 administered subcutaneously (SC) once two week for 24 weeks.
  Interventions: Drug: RAY1225
- Placebo (cohort 1) (Placebo Comparator): Participants received Placebo administered SC once two weeks for 24 weeks.
  Interventions: Drug: Placebo
- RAY1225 (cohort 2) (Experimental): Escalating doses of RAY1225 administered subcutaneously (SC) once two week
  Interventions: Drug: RAY1225
- Placebo (cohort 2) (Placebo Comparator): Participants received Placebo administered SC once two week
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RAY1225 — Administered SC
  Arms: RAY1225 (cohort 1); RAY1225 (cohort 2)
Drug: Placebo — Placebo
  Arms: Placebo (cohort 1); Placebo (cohort 2)

SUMMARY:
The main purpose of this study is to learn more about the Tolerability of RAY1225 in participants with Obesity. The study will also explore the efficacy of RAY1225. The study will last about six months for each participant.

ELIGIBILITY:
Inclusion Criteria:

1. Have a body mass index (BMI) of ≥28 kilogram per square meter (kg/m²) or ≥24 kg/m² and previously diagnosed with at least one of the following weight related comorbidities: hypertension, dyslipidemia, obstructive sleep apnea, fatty liver disease,or HbA1c ≥5.7% and < 6.5%;
2. Participants (including partners) must use reliable methods of contraception during the study and until 6 months following the last dose of investigational product.

Exclusion Criteria:

1. Obesity induced by other endocrinologic disorders or monogenetic or syndromic forms of obesity
2. with a history of diabetes or hypoglycemia;
3. Have a family or personal history of medullary thyroid carcinoma (MTC) or Multiple Endocrine Neoplasia (MEN) Syndrome type 2 or with thyroid nodules of unknown etiology found at screening and considered clinically significant by the investigator.
4. Have a prior or planned surgical treatment for obesity (excluding liposuction or abdominoplasty if performed >1 year prior to screening)
5. allergic constitution;
6. not suitable for subcutaneous injection.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Body Weight | Baseline,Week26
  Percent Change from Baseline in Body Weight

SECONDARY OUTCOMES:
Percentage of Participants Who Achieve ≥10% Body Weight Reduction | Baseline,Week26
Percentage of Participants Who Achieve ≥15% Body Weight Reduction | Baseline,Week26
Percentage of Participants Who Achieve ≥5% Body Weight Reduction | Baseline,Week26
Change from Baseline in Waist Circumference in Centimeter | Baseline,Week26

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijingcun, Hebei, China

IPD SHARING:
Plan to Share IPD: Undecided